CLINICAL TRIAL: NCT02212548
Title: Prostate-Rectal Separation With PEG Hydrogel and Its Effect on Decreasing Rectal Dose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal North Shore Hospital (Other)
Responsible Party: Principal Investigator, Professor Thomas Eade, Dr., Royal North Shore Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hydrogel
Record Dates: First submitted 2012-06-05; First posted 2014-08-08 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Cancer of the Prostate
Keywords: SpaceOAR Hydrogel Image Guided Modulated Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hydrogel (Experimental): The patient will be in the dorsal lithotomy position and prepared and draped. A transrectal ultrasound (TRUS) will be used for alignment of the needle and to ensure safe delivery. The hydrogel precursor and accelerator solutions will be mixed and connected to the Y connector that has been flushed with saline and to a syringe holder that ensures both syringe barrels are injected at the same time. After aspirating to ensure the tip of the needle is not intravascular, the perirectal space will be adequately dissected from the apex to midgland by injecting saline into the space between denonvilliers fascia and the anterior rectal space under TRUS guidance. Maintaining the needle position and angulation, the saline syringe is disconnected and the hydrogel system connected. After aspirating to ensure the needle tip is not in a blood vessel and under TRUS guidance, the 'PEG Hydrogel (SpaceOAR) is injected in a smooth, continuous technique.
  Interventions: Device: PEG Hydrogel (SpaceOAR)

INTERVENTIONS:
Device: PEG Hydrogel (SpaceOAR) — A single injection of PEG hydrogel (SpaceOAR) through the perineum under transrectal ultrasound guidance while under general anaesthetic.

SUMMARY:
This is a Phase I prospective study of 30 patients to determine whether PEG hydrogel (SpaceOAR) reduces the dose of radiation delivered to the rectum during Image Guided Intensity Modulated Radiotherapy (IG-IMRT) for prostate cancer, by increasing the space between the prostate and the rectum.

DETAILED DESCRIPTION:
Patients who are referred to the Northern Sydney Cancer Centre for radiotherapy for treatment of their prostate cancer will be screened at the initial consultation for suitability for participation in the study. Following informed consent, those who agree to participate in the study will undergo the following procedures. Blood tests will be performed to ensure normal coagulation profile and renal function prior to any procedure. Under transrectal ultrasound guidance, patients will have insertion of fiducial gold seeds into the prostate under anaesthesia. While the patient is in theatre and under anaesthesia, the PEG hydrogel (SpaceOAR) will be inserted by Dr Thomas Eade, who will be competent in the procedure. The patient will be in the dorsal lithotomy position and prepared and draped. A transrectal ultrasound (TRUS) will be used for alignment of the needle and to ensure safe delivery. The hydrogel precursor and accelerator solutions will be mixed and connected to the Y connector that has been flushed with saline and to a syringe holder that ensures both syringe barrels are injected at the same time (comes with commercial product). The solutions will be injected within 30 minutes of mixing. After aspirating to ensure the tip of the needle is not intravascular, the perirectal space will be adequately dissected from the apex to midgland by injecting saline into the space between denonvilliers fascia and the anterior rectal space under TRUS guidance. This hydrodissection, prior to delivery of the hydrogel, should create a distance of 3-4 mm between the prostate and the rectum. Maintaining the needle position and angulation, the saline syringe is disconnected and the hydrogel system connected. After aspirating to ensure the needle tip is not in a blood vessel and under TRUS guidance, the hydrogel is injected in a smooth, continuous technique. The gel sets up within approximately 8 seconds.

In order to compare the effect of the PEG hydrogel (SpaceOAR) on the dose of radiation received by the rectum, two radiotherapy plans will be created. One planning CT scan will therefore be performed prior to the injection of the PEG hydrogel and one one week following injection of the hydrogel. The two treatment plans will be created by the same radiation therapist.

As the hydrogel is clearly visible on MRI and not on CT scans, we will obtain a pelvic MRI scan following injection of the hydrogel.. The MRI scans will be used in planning and fused to the planning CT scans to aid voluming.

Treatment:

Patients will undergo standard prostate cancer planning and treatment using image guided dose escalated IMRT as per the RNSH Department protocol and guidelines to a dose of 80Gy in 40 fractions 14.

Rectal Dose Analysis:

Two plans with dose-volume histograms will be created, one using the planning CT scan from prior to the PEG hydrogel (SpaceOAR) injection and one using the planning CT and MRI performed one week post hydrogel injection. MRI scans will be obtained on the same day as the CT simulation using the same bladder filling and rectal emptying protocols. Each patient will have two plans created by the same Radiation Therapist. This will allow for comparison between the 2 plans. The patient will be treated according to the post PEG hydrogel injection plan, with the initial plan for comparison purposes only. The volume of rectum receiving 80Gy, 75Gy, 70Gy, 65Gy, 60Gy, 40Gy, 35Gy and 25Gy will be compared with the two plans.

Patient assessment:

Patients will be assessed immediately post injection of the hydrogel, 24hrs later by telephone and 1 week later by telephone to determine if there has been any adverse event related to the PEG hydrogel (SpaceOAR) injection. This will include questions regarding pain or discomfort, infection, bleeding, and changes in bowel or bladder function. Information about every adverse event will be collected and recorded on the appropriate case report form. Adverse events will be described by duration (start and end dates), severity grade, and action taken. A follow-up report will follow the initial report within 5 working days. Any reports where the adverse event has not resolved at this time will be followed up to resolution of the event or until it becomes chronic and a statement is made to this effect.

During radiotherapy treatment patients will be assessed weekly in the clinic and their toxicity will be recorded using the modified RTOG and National Cancer Institute Common Terminology Criteria (v4.0) for adverse events.

Patients will be reviewed in the clinic 3 months, 9 months, 15 months and 21 months post completion of treatment and rectal toxicity will be assessed using the modified RTOG and National Cancer Institute Common Terminology Criteria (v4.0) for adverse events.

Adverse events:

An adverse event is any undesirable experience associated with the use of a medical product in a patient. All adverse events will be appropriately reported by duration (start and end dates), severity grade, and action taken on the appropriate case report form.

Grade 1 or mild events are easily tolerated. Grade 2 or moderate events cause enough discomfort to interfere with usual activity.

Grade 3 or severe events result in inability to carry out usual activities. Grade 4 events are life threatening or disabling. The serious adverse event will be documented and medically assessed by the investigator. As the PEG hydrogel cannot be removed following injection, patients will be treated medically and symptomatically. A follow-up report will follow the initial report within 5 working days. Any reports where the adverse event has not resolved at this time will be followed up to resolution of the event or until it becomes chronic and a statement is made to this effect.

ELIGIBILITY:
Inclusion Criteria:

1. Prostate cancer, confirmed with histopathology specimen;
2. Eligible for prostate radiotherapy, either for definitive treatment or to aid local control in patients with known metastatic disease.

Exclusion criteria:

1. Metastatic disease where local radiotherapy is not recommended management
2. Complications following prostate biopsy including infection
3. Urinary retention symptoms
4. Bleeding disorder
5. Renal impairment
6. Anal fistula or perianal abscess

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
% volume of rectum receiving 40Gy, 65Gy, 70Gy, 75Gy and 80Gy | CT scans taken 1-2 weeks apart (Pre and post Hydrogel insertion)
  Estimated % volume of rectum as measured on CT dosimetry based on CT scans ore and post insertion of hydrogel taken 1-2 weeks apart (% volume of rectum receiving 40Gy, 65Gy, 70Gy, 75Gy and 80Gy).
Evaluation of serious adverse events or complications secondary to PEG hydrogel insertion. | Post-Hydrogel Insertion then 2nd weekly during radiation therapy up to 9 weeks and at a 3 month follow-up.
  Physcian reported toxicity using CTC

SECONDARY OUTCOMES:
Gastrointestinal toxicity | Second weekly evaluation during radiation therapy up to 9 weeks and at 3 mths, 9 mths, 15 mths, 21 mths, 27mths and 36mths post treatment.
  Patients will be physician scored using the CTC and patient scored using the EPIC QOL questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Eade, MD, Principal Investigator — Royal North Shore Hospital
Locations (1):
- Northern Sydney Cancer Centre, Royal North Shore Hospital, St Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Other centres with ethics approval to use annonymised data

REFERENCES:
- [Result] Juneja P, Kneebone A, Booth JT, Thwaites DI, Kaur R, Colvill E, Ng JA, Keall PJ, Eade T. Prostate motion during radiotherapy of prostate cancer patients with and without application of a hydrogel spacer: a comparative study. Radiat Oncol. 2015 Oct 24;10:215. doi: 10.1186/s13014-015-0526-1. PMID 26499473
- [Result] van Gysen K, Kneebone A, Alfieri F, Guo L, Eade T. Feasibility of and rectal dosimetry improvement with the use of SpaceOAR(R) hydrogel for dose-escalated prostate cancer radiotherapy. J Med Imaging Radiat Oncol. 2014 Aug;58(4):511-6. doi: 10.1111/1754-9485.12152. Epub 2014 Mar 3. PMID 24580893